CLINICAL TRIAL: NCT03279029
Title: Aortic Valve Regurgitation Acquired After Left Ventricular Assist Device Implantation: an Outstanding in Vivo Model of Valvular Heart Diseases
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: 2 patients included only
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2017-08; 2017-A00680-53 (Other: idrcb)
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Aortic Valve Regurgitation Acquired
MeSH Terms: interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with aortic valve disease (AVD). (Experimental)
  Interventions: Biological: blood samples; Biological: biopsy
- patients with left ventricular assist device (LVAD (Experimental)
  Interventions: Biological: blood samples; Biological: biopsy

INTERVENTIONS:
Biological: blood samples — blood samples
Biological: biopsy — biopsy of aortic valve

SUMMARY:
To investigate histological structure and molecular changes involved on the onset of AVD after left ventricular assist device (LVAD) implantation and to compare them with those of patients operated on for severe aortic regurgitation.

Methods: Bridge-to-transplant patients with AVD post-LVAD implantation are included. Patients operated on for severe aortic regurgitation are included as control. Clinical and TTE data are compiled. Samples of aortic valve are collected at the time of the intervention. RNA-sequencing analysis is performed in LVAD patients and variations of gene expression are validated by real time qPCR in both. Blood sampling are performed pre-operatively and at one-month follow up to assess the plasma level of previously identified gene modulators. In-vitro studies exposing VICs and VECs to several mechanical stimuli are performed for validation.

Conclusion(s) Taking together, the in-vivo and in-vitro models would provide important information for the understanding of valve remodeling and disease. ECM gene modulators could represent pertinent molecular targets to stop the progression of AVD

ELIGIBILITY:
Inclusion Criteria:

* Patients with long-term left-ventricular assistance awaiting transplant
* Patients with severe aortic surgical spring deficiency
* Major Patient

Exclusion Criteria:

* Minor Patient
* Pregnant or nursing women
* Major under guardianship
* People in emergencies
* Persons not covered by the social security scheme

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2017-09-14 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2023-08-08 (Estimated)

PRIMARY OUTCOMES:
blood sample | 24 months
  RNA-sequencing analysis

CONTACTS AND LOCATIONS:
Overall Officials: alexis THERON, Principal Investigator — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France